CLINICAL TRIAL: NCT04451122
Title: Treatment of Ocular Demodicosis by Cleansing the Eyelid Margins Combined With Tea Tree Oil Ointment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, Researcher；clinical research center, Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: demodicosis WDD
Record Dates: First submitted 2020-04-16; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Mite-Borne
Keywords: eyelid margins; ocular demodicosis
MeSH Terms: interventions — Tea Tree Oil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of ocular demodicosis (Other)
  Interventions: Other: cleansing the eyelid margins

INTERVENTIONS:
Other: cleansing the eyelid margins — using eyelid cleaning wipes to cleansing the eyelid margins
  Other Names: tea tree oil

SUMMARY:
To investigate whether the cleaning of eyelid margins increases the effectiveness of traditional tea tree oil eyelid margins in treating mites. The investigators randomly divided 60 participants into two groups: Group A was treated with traditional tea tree oil eyelid margin, Group B was treated with traditional tea tree oil eyelid margin + eyelid cleansing, and participants were rechecked after 3 months of regular medication.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosisof ocular surface mite parasitism

Exclusion Criteria:

* any acute keratoconjunctivitis;c dacryocystitis

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
The severity of dry eyes | 3 months
  OSDI dry eye questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China